CLINICAL TRIAL: NCT02667899
Title: The Consciousness Variation of Deep Brain Stimulation (DBS) and Transcranial Magnetic Stimulation (TMS) for Disorders of Consciousness(DOC) Patients in a Large Scale Randomised Trial
Brief Title: The Consciousness Variation of Deep Brain and Transcranial Magnetic Stimulation for Disorders of Consciousness Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuehai Wu (Other)
Responsible Party: Sponsor-Investigator, Xuehai Wu, Associate Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shwuxuehai
Record Dates: First submitted 2015-12-20; First posted 2016-01-29 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Consciousness Disorders
Keywords: disorders of consciousness; deep brain stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Consciousness Disorders | interventions — Deep Brain Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DBS group (Active Comparator): Besides routine treatment, Doc patients in this group will accepted deep brain stimulation treatment.
  Interventions: Device: deep brain stimulation
- TMS group (Active Comparator): Besides routine treatment, Doc patients in this group will accepted transcranial magnetic stimulation treatment.
  Interventions: Device: transcranial magnetic stimulation
- Control group (Placebo Comparator): This Doc patients will accepted routine treatment.
  Interventions: Other: Routine treatment

INTERVENTIONS:
Device: deep brain stimulation — Deep brain stimulation means stimulate the brain with DBS.
  Arms: DBS group
Device: transcranial magnetic stimulation — Transcranial magnetic stimulation means stimulate the brain with magnetic stimulation.
  Arms: TMS group
Other: Routine treatment — Means without above additional treatment.
  Arms: Control group

SUMMARY:
Aims:To explore the consciousness stimulation role of DBS (Deep Brain Stimulation) and TMS (Transcranial Magnetic Simulation) for DOC (Disorders of Consciousness) patients.

Methods:Seventy-five DOC patients will be randomised into three groups: DBS group, TMS group and Control group. Three months after treatments, the result will be analysed and concluded.

DETAILED DESCRIPTION:
To explore the consciousness stimulation role of DBS (Deep Brain Stimulation) and TMS (Transcranial Magnetic Stimulation) for DOC (Disorders of Consciousness) patients. Seventy-five DOC patients will be randomised into three groups: DBS group, TMS group and Control group. These patients will be recorded the conscious level, fMRI (functional magnetic resonance imaging) and EEG evaluation before treatment of research, and three months later the prognosis was also recorded. Finally, the variation of consciousness, prognosis, fMRI and EEG index for three groups will be analyzed and compared. Hopefully, there will be a conclusion for these treatments to DOC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 14 to 65 years old;
2. DOC patients, including vegetative state and minimally consciousness state.
3. With normal body temperature, stable vital signs, spontaneous breathing without extra oxygen supply, no tracheotomy using metal trachea cannula, and feasible for magnetic resonance inspectors;
4. Written informed consent from patient families

Exclusion Criteria:

1. History with nervous or spirit disorders, or some other serious diseases such as cardiac or pulmonary problems;
2. Patients with V-P shunt or ommaya implantation, which may effects magnetic resonance scan signal analysis;
3. Body temperature is abnormal, vital signs is not stable, still need ventilator to support breathing; Plentiful sputum needed suction during MRI scans.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
The consciousness variation of DBS and TMS for DOC Patients in a large scale randomised trial (revised-coma recovery scale) | 3 months
  revised-coma recovery scale(CRS-R)

SECONDARY OUTCOMES:
The conscious index based on fMRI | 3 months
  Using fMRI to evaluate consciousness in DoC patients
The conscious index based on EEG | 3 months
  Using EEG to evaluate consciousness in DoC patients

CONTACTS AND LOCATIONS:
Overall Officials: Xuehai Wu, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Department of Neurosurgery, Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Ok. All participant data which can be shared will include these patient's clinical information, consciousness level and prognosis scores. Who want to share data can email to our group for data and we will glad to share.